CLINICAL TRIAL: NCT04122092
Title: Application of Ultrasensitive Chromosomal Aneuploidy Detection (UCAD) as a Surrogate Biomarker of Minimal Residual Diseases for Multiple Myeloma Patients
Brief Title: Evaluation of Ultrasensitive Chromosomal Aneuploidy Detection for Detecting Minimal Residual Disease in Multiple Myeloma
Acronym: EUCADD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Juan Du, Deputy director of hematology, Shanghai Changzheng Hospital
Other Study IDs: cz-pg001
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Minimal residual disease; Chromosomal aneuploidy detection; Chromosomal instability
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual; Chromosomal Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood were collected from MM patients satisfied cohort condition and stored in cell-free DNA-protectant immediately after collection. Cell-free DNA from peripheral blood will be analyzed by Ultrasensitive Chromosomal Aneuploidy Detection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MM patients have curative effect at least VGPR: We will detect cfDNA CIN of multiple myeloma patients who have the curative effect at least very good partial response (VGPR) after front line therapy, and then monitoring cfDNA CIN every two treatment cycles or every three months during follow up，the result will be compared with bone marrow aspiration MFC.
  Interventions: Diagnostic Test: The level of plasma cfDNA CINs

INTERVENTIONS:
Diagnostic Test: The level of plasma cfDNA CINs — The extracted cfDNA from PB will be analyzed by UCAD to determine the level of CINs

SUMMARY:
Despite the significantly higher complete remission rates and improved survival achieved over the last decade，multiple myeloma (MM) patients continue to relapse due to persistence of minimal residual disease (MRD). Currently, numerous studies have evaluated the prognostic value of MRD by detecting immunophenotypic and immunoglobulin (Ig) gene rearrangements from bone marrow aspiration samples. Here the investigators intend to study the clinical utility of Ultrasensitive Chromosomal Aneuploidy Detection (UCAD) as an MRD assay, which is based on plasma cell-free DNA(cfDNA) low-coverage whole-genome sequencing. UCAD is non-invasive and applicable for tumors with high heterogeneity and extramedullary invasions.

DETAILED DESCRIPTION:
In multiple myeloma, Minimal Residual Disease (MRD) refers to myeloma cells that are present in the bone marrow after a clinical response has been measured and the patient is in remission. A patient who tests "MRD negative" after treatment for myeloma has less than one myeloma cell per million bone marrow cells. Data from recent clinical trials suggest that patients with such a low level of disease may be less likely to experience a relapse of their condition than patients with higher levels. In recent years, MRD testing is now be applied in the management of patients receiving standard therapies for the disease.

Chromosomal instability(CIN) results from errors in chromosome segregation during mitosis, leading to structural and numerical chromosomal abnormalities. It will generate genomic heterogeneity that acts as a substrate for natural selection. Furthermore, it is proved that tumors with aneuploidies and polyploidy resulting from whole-genome doubling are related with metastasis, treatment resistance, and decreased overall survival. It is estimated that 60%-80% of human tumors exhibit chromosomal abnormalities suggestive of CIN. CIN positively correlates with tumor stage and is enriched in relapsed as well as metastatic tumor specimens. Due to the ubiquity of CIN in cancer cells and cancer cell releasing DNA into peripheral blood (PB) when apoptosis, it is a potentially non-invasive way to detect CIN in PB cfDNA from the MM patients to character MRD level. UCAD is a new method to detecting CIN in the DNA sample from patients, including extracting cfDNA from PB, analyzing DNA by low-coverage whole-genome sequencing, processing the data by bio-information techniques, and finally optimizing the management of MM patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients new diagnosed with MM and with the curative effect at least VGPR.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years
* Individuals unwilling to sign the consent form or unwilling to provide PB for test or unwilling to provide the medical record.
* Individuals unwilling to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with MM and with the curative effect at least VGPR in Changzheng Hospital from Aug 2019 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of the prognostic of the MRD negative and MRD positive defined by UCAD | 36month
  The patients' prognostic was evaluated with the median time of progress free survival (PFS) and overall survival (OS)
The concordance rate analysis between UCAD and multiparameter flow cytometry(MFC) | 36month
  number of patients "declared MRD positive or MRD negative" with the UCAD and MFC test simultaneously among the patients being tested successfully with both

SECONDARY OUTCOMES:
The applicability analysis of UCAD | 36month
  number of patients being tested successfully with the UCAD among the patients included in this cohort
The MRD negative rate analysis among VGPR patients | 24month
  The MRD negative patients accounted for the total enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Du, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakhoum SF, Ngo B, Laughney AM, Cavallo JA, Murphy CJ, Ly P, Shah P, Sriram RK, Watkins TBK, Taunk NK, Duran M, Pauli C, Shaw C, Chadalavada K, Rajasekhar VK, Genovese G, Venkatesan S, Birkbak NJ, McGranahan N, Lundquist M, LaPlant Q, Healey JH, Elemento O, Chung CH, Lee NY, Imielenski M, Nanjangud G, Pe'er D, Cleveland DW, Powell SN, Lammerding J, Swanton C, Cantley LC. Chromosomal instability drives metastasis through a cytosolic DNA response. Nature. 2018 Jan 25;553(7689):467-472. doi: 10.1038/nature25432. Epub 2018 Jan 17. PMID 29342134
- [Background] Hieronymus H, Murali R, Tin A, Yadav K, Abida W, Moller H, Berney D, Scher H, Carver B, Scardino P, Schultz N, Taylor B, Vickers A, Cuzick J, Sawyers CL. Tumor copy number alteration burden is a pan-cancer prognostic factor associated with recurrence and death. Elife. 2018 Sep 4;7:e37294. doi: 10.7554/eLife.37294. PMID 30178746
- [Background] Bai Y, Orfao A, Chim CS. Molecular detection of minimal residual disease in multiple myeloma. Br J Haematol. 2018 Apr;181(1):11-26. doi: 10.1111/bjh.15075. Epub 2017 Dec 19. PMID 29265356
- [Background] Martinez-Lopez J, Lahuerta JJ, Pepin F, Gonzalez M, Barrio S, Ayala R, Puig N, Montalban MA, Paiva B, Weng L, Jimenez C, Sopena M, Moorhead M, Cedena T, Rapado I, Mateos MV, Rosinol L, Oriol A, Blanchard MJ, Martinez R, Blade J, San Miguel J, Faham M, Garcia-Sanz R. Prognostic value of deep sequencing method for minimal residual disease detection in multiple myeloma. Blood. 2014 May 15;123(20):3073-9. doi: 10.1182/blood-2014-01-550020. Epub 2014 Mar 19. PMID 24646471
- [Background] Oberle A, Brandt A, Voigtlaender M, Thiele B, Radloff J, Schulenkorf A, Alawi M, Akyuz N, Marz M, Ford CT, Krohn-Grimberghe A, Binder M. Monitoring multiple myeloma by next-generation sequencing of V(D)J rearrangements from circulating myeloma cells and cell-free myeloma DNA. Haematologica. 2017 Jun;102(6):1105-1111. doi: 10.3324/haematol.2016.161414. Epub 2017 Feb 9. PMID 28183851
- [Background] Rihova L, Vsianska P, Bezdekova R, Kralova R, Penka M, Krejci M, Pour L, Hajek R. Minimal Residual Disease Assessment in Multiple Myeloma by Multiparametric Flow Cytometry. Klin Onkol. 2017 Summer;30(Supplementum2):21-28. doi: 10.14735/amko20172S21. PMID 28903567
- [Background] Berger N, Kim-Schulze S, Parekh S. Minimal Residual Disease in Multiple Myeloma: Impact on Response Assessment, Prognosis and Tumor Heterogeneity. Adv Exp Med Biol. 2018;1100:141-159. doi: 10.1007/978-3-319-97746-1_9. PMID 30411265
- [Background] Li H, Li F, Zhou X, Mei J, Song P, An Z, Zhao Q, Guo X, Wang X, Zhai Y. Achieving minimal residual disease-negative by multiparameter flow cytometry may ameliorate a poor prognosis in MM patients with high-risk cytogenetics: a retrospective single-center analysis. Ann Hematol. 2019 May;98(5):1185-1195. doi: 10.1007/s00277-019-03609-x. Epub 2019 Feb 5. PMID 30721336